CLINICAL TRIAL: NCT07264413
Title: Bleeding Reduction in Grade II-III Haemorrhoids Through Embolization Treatment
Acronym: BRIGHT
Status: Not yet recruiting | Type: Observational
Sponsor: Cardiovascular and Interventional Radiological Society of Europe (Other)
Collaborators: Medtronic (Industry); Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: BRIGHT
Record Dates: First submitted 2025-11-20; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hemorrhoid; Hemorrhoid Bleeding
Keywords: Haemorrhoids; Grade II-III haemorrhoids; Symptomatic haemorrhoids; Hemorrhoidal bleeding; Haemorrhoidal disease; Haemorrhoid artery embolization; HAE; Artery embolization; Transarterial embolization; Minimally invasive; Embolization coils
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with bleeding grade II-III haemorrhoids: Adult patients with bleeding grade II-III haemorrhoids planned to be treated with Haemorrhoid artery embolization (HAE) using embolization coils
  Interventions: Procedure: Haemorrhoid artery embolizsation (HAE)

INTERVENTIONS:
Procedure: Haemorrhoid artery embolizsation (HAE) — Haemorrhoid artery embolization (HAE) is a minimally invasive procedure used to treat symptomatic haemorrhoids by reducing their blood supply. Under imaging guidance, typically fluoroscopy, a catheter is inserted through a small puncture in the groin or wrist and guided into the arteries that supply the haemorrhoidal tissue, known as the superior rectal arteries.
  Once the target vessels are identified, embolization coils-tiny metal coils designed to block blood flow-are placed inside these arteries. The coils create a controlled blockage, decreasing blood flow to the haemorrhoids, which helps shrink the swollen tissue and reduce bleeding.
  HAE is usually performed as an day-case procedure under local anaesthesia with mild sedation, and tends to result in less pain, quicker recovery, and lower complication rates compared to surgical approaches.
  Other Names: Embolization Coils

SUMMARY:
BRIGHT is a Europe-wide study that will follow up to 250 adults with bleeding symptoms from haemmorhoids (Grade II-III categories). It aims to understand how well a minimally invasive procedure called haemorrhoid artery embolization (HAE) works in everyday clinical practice, which is a technique that blocks the blood vessels feeding the haemorrhoids. As this technique does not require major surgery, HAE offers several benefits such as less trauma, quicker recovery, and the use of only local anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients presenting bleeding Grade II-III haemorrhoids with French bleeding score ≥3 planned to be treated with HAE using embolization coils;
2. Patients competent and willing to give written informed consent.

Exclusion Criteria:

1. Minors and other vulnerable populations who may not be able to give informed consent freely or for whom participation is not essential to the study (incapacitated and unconscious individuals, persons deprived of liberty, pregnant and breastfeeding women, etc.);
2. Patients receiving HAE using a combination of coils and particles, particles only, or any other embolic agents;
3. Patients who have had previous surgical haemorrhoidectomy at any time or other treatments for haemorrhoids within 1 year before the planned HAE;
4. Patients with known perianal sepsis, inflammatory bowel disease, peri-anal fistula, colorectal malignancy or pre-existing sphincter injury resulting in incontinence;
5. Patients with an immunodeficiency;
6. Known severe atheromatous disease with occlusion of target vessels preventing embolization;
7. Absolute contraindication to contrast media;
8. ECOG performance status > 2;
9. Life expectancy < 12 months;
10. Patients with unstable angina;
11. Patients currently taking nicorandil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with bleeding grade II-III haemorrhoids (French Bleeding Score ≥3) planned to be treated with HAE coil-only embolization who fit the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Haemorrhoidal bleeding | 12 months
  Evaluated using the French Bleeding Score.

SECONDARY OUTCOMES:
Haemorrhoidal bleeding | 1, 3 and 24 months
  Evaluation of haemorrhoidal bleeding at time points listed below compared to baseline using the French Bleeding Score.
Patient-reported Pain using the Visual Analogue Scale | 1 day, 1- and 3-months post treatment, compared to baseline
  The 10 cm Visual Analogue Scale (VAS) is a patient-reported outcome measure used to assess the intensity of a symptom such as pain, discomfort, or bleeding. It consists of a straight, 10-centimeter horizontal line with two anchored endpoints: 0 cm = no symptom, and 10 cm = worst imaginable symptom. Participants mark a point on the line that best represents the severity of their symptom at the time of assessment. This will be measured at 1 day, 1- and 3-months after the treatment.
Patient-reported Pain measured by Analgesic intake | 1 day, 1- and 3-months post treatment
  Analgesic intake refers to the use of any pain-relief medication taken to manage haemorrhoid-related discomfort after HAE. This includes over-the-counter or prescribed agents such as acetaminophen/paracetamol or NSAIDs. Participants will be recorded as having taken analgesics if they use any pain medication for haemorrhoid symptoms during the specified time frame.
Frequency and severity of procedural complications and other adverse events | Within 3 months after the HAE procedure
  The severity of complications and procedure-related adverse events will be graded according to the Clavian Dindo classification system.
Functional recovery | From the procedure date until the patient returns to work or usual daily activities (Number of days)
  Measured as the number of days until the patient is fit enough to return to work or other usual daily activities.
Freedom from recurrence | 1, 3, 12 and 24 months
  Defined as the proportion of patients with cured or improved symptoms as described in the HubBle Trial.
Clinical appearance of haemorrhoids | 12 months
  Evaluated at proctoscopy at 12 months if done per SOC or following recurrence requiring further intervention.
Patient-reported symptoms | 3, 12 and 24 months
  Evaluated using the Haemorrhoids Severity Score at the specified time points below compared to baseline.
Patient-reported continence | 3 months
  Assessed using the Vaizey Incontinence Score at the specified time points below compared to baseline.
Patient-reported health-related quality-of-life | 1 day, 1-, 3-, 12- and 24-months
  Measured by EuroQol Five-Dimension, Five-Level Questionnaire (EuroQol EQ-5D-5L) at the specified time points below compared to baseline. It is a standardized, participant-reported measure of health-related quality of life that assesses five dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-each rated on five levels of severity: no problems, slight problems, moderate problems, severe problems, and extreme problems/unable to perform. Higher EQ-5D-5L index values indicate better overall health status, while lower scores reflect poorer health, greater symptom burden, or more functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Bent, Dr, Study Chair — Royal Bournemouth Hospital, University Hospitals Dorset NHS Foundation Trust; Christoph A. Binkert, Prof. Dr. med., Study Chair — Medical Radiological Institute; Roberto Iezzi, Prof., Study Chair — Fondazione Policlinico Agostino Gemelli, IRCCS Catholic University; Vincent Vidal, Prof., Study Chair — Marseille University Hospital Timone

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown SR, Tiernan JP, Watson AJM, Biggs K, Shephard N, Wailoo AJ, Bradburn M, Alshreef A, Hind D; HubBLe Study team. Haemorrhoidal artery ligation versus rubber band ligation for the management of symptomatic second-degree and third-degree haemorrhoids (HubBLe): a multicentre, open-label, randomised controlled trial. Lancet. 2016 Jul 23;388(10042):356-364. doi: 10.1016/S0140-6736(16)30584-0. Epub 2016 May 25. PMID 27236344
- [Background] Vaizey CJ, Carapeti E, Cahill JA, Kamm MA. Prospective comparison of faecal incontinence grading systems. Gut. 1999 Jan;44(1):77-80. doi: 10.1136/gut.44.1.77. PMID 9862829
- [Background] Nystrom PO, Qvist N, Raahave D, Lindsey I, Mortensen N; Stapled or Open Pile Procedure (STOPP) trial study group. Randomized clinical trial of symptom control after stapled anopexy or diathermy excision for haemorrhoid prolapse. Br J Surg. 2010 Feb;97(2):167-76. doi: 10.1002/bjs.6804. PMID 20035531
- [Background] Fathallah N, Beaussier H, Chatellier G, Meyer J, Sapoval M, Moussa N, de Parades V. Proposal for a New Score: Hemorrhoidal Bleeding Score. Ann Coloproctol. 2021 Oct;37(5):311-317. doi: 10.3393/ac.2020.08.19. Epub 2020 Sep 18. PMID 32972102
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542